CLINICAL TRIAL: NCT06714227
Title: Genetics of Prostate Cancer in Young Patients
Acronym: ProK55
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ProK55; RC 2022-2024 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-11-28; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Peripheral blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with prostate carcinoma before the age of 55: Exome sequencing (WES) of genomic DNA
  Interventions: Genetic: Molecular analysis of genomic DNA (exome sequencing) from peripheral blood sample

INTERVENTIONS:
Genetic: Molecular analysis of genomic DNA (exome sequencing) from peripheral blood sample — The first level of investigation will focus on genes already described in cases of pathogenic germline variants of prostate cancer and/or DNA repair system genes. The second level of investigation will consider variants in genes known to confer increased risk of cancer development, e.g., genes listed in the UK health system's solid tumor predisposition gene panel. Finally, pathogenic/probably pathogenic variants in the exome in genes attributable to increased risk will be evaluated on the basis of molecular pathway and findings in the scientific literature.

SUMMARY:
The aim of the study is to identify genetic variants in genes responsible or potentially responsible for the etiology of prostate cancer in a population of patients with early onset of the malignancy.

DETAILED DESCRIPTION:
The data collected from the study will provide a preliminary picture of the prevalence and type of germline pathological variants in the context of early-onset prostate cancer in the Italian population. In addition, alterations in DNA repair genes other than BRCA1-2 and ATM, including any genes yet undescribed as causative or predisposing, have yet to be explored in detail: in many cases the significance of variants is not well defined in terms of pathogenicity, prognostic value, and predictive indicator of response to different treatments. Therefore, an extensive mutational analysis-even if performed on a limited number of patients-can generate a large number of variants for evaluation, bringing knowledge about the relationship between these variants and the onset of malignancy The information obtained, although merely exploratory, may indicate the desirability of conducting systematic genetic investigations in this particular patient population in the future, especially in view of the new therapeutic strategies available such as immunotherapy or PARP inhibitors

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic or cytologic diagnosis of prostate cancer
* Age ≥18 years and ≤55 years at first diagnosis of prostate carcinoma
* Availability of clinical and instrumental data related to prostate cancer
* Patients who knowingly express willingness to participate in the study after signing written informed consent

Exclusion Criteria:

* None

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of patients aged 18 years or older with a diagnosis of prostate cancer and age ≤55 years at first diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Presence/absence and type of pathogenic/probably pathogenic germline variants in genes previously implicated in prostate cancer etiology | 4 years
  molecular analysis of genomic DNA

SECONDARY OUTCOMES:
Presence/absence and type of variants in genes potentially implicated in the etiology of prostate cancer (candidate genes). | 4 years
  molecular analysis of genomic DNA

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Rossi, Biologist, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
IPD not included in the protocol approved by the ethics committee